CLINICAL TRIAL: NCT04043286
Title: The Effects of Disconnection and Reconnection of Definitive Abutments on Peri-Implant Bone Levels: A 1-year Split-Mouth Randomized Controlled Clinical Study
Brief Title: The Effects of Dis/Reconnection of Implant Abutments on Peri-implant Bone Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: Nobel Biocare (Industry)
Responsible Party: Principal Investigator, Joseph Kan, DDS, Professor, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5190024
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Results first posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Bone Loss; Implant Complication; Gingival Recession
Keywords: One abutment one time; Disconnection and reconnection; Definitive abutment
MeSH Terms: conditions — Bone Diseases, Metabolic; Gingival Recession

STUDY DESIGN:
Intervention Model Description: Single center, prospective, randomized modified split mouth clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control group (No Intervention): Split mouth: Healing abutments are connected on the implants on the day of surgery, which will be subjected to multiple disconnection and reconnection during the study
- Test group (Experimental): Split mouth: Definitive abutments connected to the implants on the day of surgery. No disconnection or reconnection during the prosthetic phase
  Interventions: Device: Definitive abutment

INTERVENTIONS:
Device: Definitive abutment — With two height options available, On1 Base are selected depending on the thickness of the soft tissue. It remains in position from implant placement to finalization, which leaves the soft tissue undisturbed for optimized healing, moved the restorative platform of Nobel Biocare conical connection implants from bone level to tissue level, thereby simplifying the restorative procedures
  Other Names: On1 Base; On1 Concept
  Arms: Test group

SUMMARY:
The aim of this study was to evaluate the effects of definitive abutment connection at the time of implant placement on peri-implant bone levels and soft tissue changes in posterior maxilla and mandible regions.

DETAILED DESCRIPTION:
A total of 38 implants were placed in 17 patients with at least 2 missing posterior teeth in the maxilla or the mandible for this study. Each patient received 2 or 4 implants. A definitive prefabricated abutment (test group) was randomly connected to one implant at implant placement (T0) and left undisturbed throughout the duration of the study. On the other implant, a healing abutment (control group) was connected and subjected to go through three disconnections and reconnections at 3 months (T3), 6 months (T6), and 12 months (T12) after the implant placement. Throughout the study period (1 year), all implants remained unrestored. Marginal bone level changes (MBLC) were assessed using standardized periapical radiographs taken at T0 and T12. Peri-implant soft tissue parameters including the keratinized mucosa width and lingual mucosa thickness were also recorded and evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age 18
* Good oral hygiene
* Healed site that possess two or more missing teeth in the maxillary or mandibular posterior region (excluding third molars)
* Adequate bone to accommodate at least a 4.3 mm diameter and 8mm length implant at each site
* Have at least 8mm interocclusal restorative space
* Willing to participate and attend the planned follow-up visits.

Exclusion Criteria:

* History of alcohol/drug dependency, or any medical, physical, or psychological factor that might affect the surgical or prosthodontic procedures and follow-up examinations
* History of radiation therapy to the head and neck region
* History or current habit of smoking
* History or current habit of bruxism
* No opposing occluding dentition or prostheses
* Need for bone augmentation during implant placement
* Implant insertion torque value <35 Ncm

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Kan, DDS, MS, Principal Investigator — Loma Linda University School of Dentistry
Locations (1):
- Loma Linda University, School of Dentistry, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abrahamsson I, Berglundh T, Wennstrom J, Lindhe J. The peri-implant hard and soft tissues at different implant systems. A comparative study in the dog. Clin Oral Implants Res. 1996 Sep;7(3):212-9. doi: 10.1034/j.1600-0501.1996.070303.x. PMID 9151585
- [Background] Berglundh T, Lindhe J, Ericsson I, Marinello CP, Liljenberg B, Thomsen P. The soft tissue barrier at implants and teeth. Clin Oral Implants Res. 1991 Apr-Jun;2(2):81-90. doi: 10.1034/j.1600-0501.1991.020206.x. PMID 1809403
- [Background] Berglundh T, Lindhe J. Dimension of the periimplant mucosa. Biological width revisited. J Clin Periodontol. 1996 Oct;23(10):971-3. doi: 10.1111/j.1600-051x.1996.tb00520.x. PMID 8915028
- [Background] Squier CA, Collins P. The relationship between soft tissue attachment, epithelial downgrowth and surface porosity. J Periodontal Res. 1981 Jul;16(4):434-40. doi: 10.1111/j.1600-0765.1981.tb00994.x. No abstract available. PMID 6459440
- [Background] Chehroudi B, Gould TR, Brunette DM. The role of connective tissue in inhibiting epithelial downgrowth on titanium-coated percutaneous implants. J Biomed Mater Res. 1992 Apr;26(4):493-515. doi: 10.1002/jbm.820260407. PMID 1601902
- [Background] Ericsson I, Persson LG, Berglundh T, Marinello CP, Lindhe J, Klinge B. Different types of inflammatory reactions in peri-implant soft tissues. J Clin Periodontol. 1995 Mar;22(3):255-61. doi: 10.1111/j.1600-051x.1995.tb00143.x. PMID 7790533
- [Background] Broggini N, McManus LM, Hermann JS, Medina RU, Oates TW, Schenk RK, Buser D, Mellonig JT, Cochran DL. Persistent acute inflammation at the implant-abutment interface. J Dent Res. 2003 Mar;82(3):232-7. doi: 10.1177/154405910308200316. PMID 12598555
- [Background] Rompen E. The impact of the type and configuration of abutments and their (repeated) removal on the attachment level and marginal bone. Eur J Oral Implantol. 2012;5 Suppl:S83-90. PMID 22834397
- [Background] Abrahamsson I, Berglundh T, Lindhe J. The mucosal barrier following abutment dis/reconnection. An experimental study in dogs. J Clin Periodontol. 1997 Aug;24(8):568-72. doi: 10.1111/j.1600-051x.1997.tb00230.x. PMID 9266344
- [Background] Becker K, Mihatovic I, Golubovic V, Schwarz F. Impact of abutment material and dis-/re-connection on soft and hard tissue changes at implants with platform-switching. J Clin Periodontol. 2012 Aug;39(8):774-80. doi: 10.1111/j.1600-051X.2012.01911.x. Epub 2012 Jun 7. PMID 22676071
- [Background] Rodriguez X, Vela X, Mendez V, Segala M, Calvo-Guirado JL, Tarnow DP. The effect of abutment dis/reconnections on peri-implant bone resorption: a radiologic study of platform-switched and non-platform-switched implants placed in animals. Clin Oral Implants Res. 2013 Mar;24(3):305-11. doi: 10.1111/j.1600-0501.2011.02317.x. Epub 2011 Oct 3. PMID 22092773
- [Background] Alves CC, Munoz F, Cantalapiedra A, Ramos I, Neves M, Blanco J. Marginal bone and soft tissue behavior following platform switching abutment connection/disconnection--a dog model study. Clin Oral Implants Res. 2015 Sep;26(9):983-91. doi: 10.1111/clr.12385. Epub 2014 Apr 16. PMID 24735458
- [Background] Degidi M, Nardi D, Piattelli A. One abutment at one time: non-removal of an immediate abutment and its effect on bone healing around subcrestal tapered implants. Clin Oral Implants Res. 2011 Nov;22(11):1303-7. doi: 10.1111/j.1600-0501.2010.02111.x. Epub 2011 Feb 24. PMID 21985288
- [Background] Degidi M, Nardi D, Daprile G, Piattelli A. Nonremoval of immediate abutments in cases involving subcrestally placed postextractive tapered single implants: a randomized controlled clinical study. Clin Implant Dent Relat Res. 2014 Dec;16(6):794-805. doi: 10.1111/cid.12051. Epub 2013 Mar 4. PMID 23458566
- [Background] Canullo L, Bignozzi I, Cocchetto R, Cristalli MP, Iannello G. Immediate positioning of a definitive abutment versus repeated abutment replacements in post-extractive implants: 3-year follow-up of a randomised multicentre clinical trial. Eur J Oral Implantol. 2010 Winter;3(4):285-96. PMID 21180681
- [Background] Grandi T, Guazzi P, Samarani R, Garuti G. Immediate positioning of definitive abutments versus repeated abutment replacements in immediately loaded implants: effects on bone healing at the 1-year follow-up of a multicentre randomised controlled trial. Eur J Oral Implantol. 2012 Spring;5(1):9-16. PMID 22518376
- [Background] Berberi AN, Sabbagh JM, Aboushelib MN, Noujeim ZF, Salameh ZA. A 5-year comparison of marginal bone level following immediate loading of single-tooth implants placed in healed alveolar ridges and extraction sockets in the maxilla. Front Physiol. 2014 Jan 31;5:29. doi: 10.3389/fphys.2014.00029. eCollection 2014. PMID 24550840
- [Background] Grandi T, Guazzi P, Samarani R, Maghaireh H, Grandi G. One abutment-one time versus a provisional abutment in immediately loaded post-extractive single implants: a 1-year follow-up of a multicentre randomised controlled trial. Eur J Oral Implantol. 2014 Summer;7(2):141-9. PMID 24977249
- [Background] Molina A, Sanz-Sanchez I, Martin C, Blanco J, Sanz M. The effect of one-time abutment placement on interproximal bone levels and peri-implant soft tissues: a prospective randomized clinical trial. Clin Oral Implants Res. 2017 Apr;28(4):443-452. doi: 10.1111/clr.12818. Epub 2016 Mar 25. PMID 27016157
- [Background] Koutouzis T, Koutouzis G, Gadalla H, Neiva R. The effect of healing abutment reconnection and disconnection on soft and hard peri-implant tissues: a short-term randomized controlled clinical trial. Int J Oral Maxillofac Implants. 2013 May-Jun;28(3):807-14. doi: 10.11607/jomi.3022. PMID 23748313
- [Background] Luongo G, Bressan E, Grusovin MG, d'Avenia F, Neumann K, Sbricoli L, Esposito M. Do repeated changes of abutments have any influence on the stability of peri-implant tissues? Four-month post-loading preliminary results from a multicentre randomised controlled trial. Eur J Oral Implantol. 2015 Summer;8(2):129-40. PMID 26021224
- [Background] Iglhaut G, Schwarz F, Winter RR, Mihatovic I, Stimmelmayr M, Schliephake H. Epithelial attachment and downgrowth on dental implant abutments--a comprehensive review. J Esthet Restor Dent. 2014 Sep-Oct;26(5):324-31. doi: 10.1111/jerd.12097. Epub 2014 Mar 11. PMID 24612047
- [Background] Smith DE, Zarb GA. Criteria for success of osseointegrated endosseous implants. J Prosthet Dent. 1989 Nov;62(5):567-72. doi: 10.1016/0022-3913(89)90081-4. PMID 2691661
- [Background] Mombelli A, van Oosten MA, Schurch E Jr, Land NP. The microbiota associated with successful or failing osseointegrated titanium implants. Oral Microbiol Immunol. 1987 Dec;2(4):145-51. doi: 10.1111/j.1399-302x.1987.tb00298.x. No abstract available. PMID 3507627
- [Background] Linkevicius T, Apse P, Grybauskas S, Puisys A. The influence of soft tissue thickness on crestal bone changes around implants: a 1-year prospective controlled clinical trial. Int J Oral Maxillofac Implants. 2009 Jul-Aug;24(4):712-9. PMID 19885413
- [Background] Wennstrom JL, Bengazi F, Lekholm U. The influence of the masticatory mucosa on the peri-implant soft tissue condition. Clin Oral Implants Res. 1994 Mar;5(1):1-8. doi: 10.1034/j.1600-0501.1994.050101.x. PMID 8038340
- [Background] Puisys A, Linkevicius T. The influence of mucosal tissue thickening on crestal bone stability around bone-level implants. A prospective controlled clinical trial. Clin Oral Implants Res. 2015 Feb;26(2):123-9. doi: 10.1111/clr.12301. Epub 2013 Dec 9. PMID 24313250
- [Background] Schwarz F, Alcoforado G, Nelson K, Schaer A, Taylor T, Beuer F, Strietzel FP. Impact of implant-abutment connection, positioning of the machined collar/microgap, and platform switching on crestal bone level changes. Camlog Foundation Consensus Report. Clin Oral Implants Res. 2014 Nov;25(11):1301-1303. doi: 10.1111/clr.12269. Epub 2013 Oct 21. PMID 24147913
- [Background] Schwarz F, Hegewald A, Becker J. Impact of implant-abutment connection and positioning of the machined collar/microgap on crestal bone level changes: a systematic review. Clin Oral Implants Res. 2014 Apr;25(4):417-25. doi: 10.1111/clr.12215. Epub 2013 Jun 18. PMID 23782338
- [Background] Schwarz F, Mihatovic I, Ferrari D, Wieland M, Becker J. Influence of frequent clinical probing during the healing phase on healthy peri-implant soft tissue formed at different titanium implant surfaces: a histomorphometrical study in dogs. J Clin Periodontol. 2010 Jun;37(6):551-62. doi: 10.1111/j.1600-051X.2010.01568.x. PMID 20507379
- [Background] Schwarz F, Mihatovic I, Golubovich V, Schar A, Sager M, Becker J. Impact of abutment microstructure and insertion depth on crestal bone changes at nonsubmerged titanium implants with platform switch. Clin Oral Implants Res. 2015 Mar;26(3):287-92. doi: 10.1111/clr.12478. Epub 2014 Aug 30. PMID 25175742
- [Background] Abrahamsson I, Berglundh T, Glantz PO, Lindhe J. The mucosal attachment at different abutments. An experimental study in dogs. J Clin Periodontol. 1998 Sep;25(9):721-7. doi: 10.1111/j.1600-051x.1998.tb02513.x. PMID 9763327
- [Background] Welander M, Abrahamsson I, Berglundh T. The mucosal barrier at implant abutments of different materials. Clin Oral Implants Res. 2008 Jul;19(7):635-41. doi: 10.1111/j.1600-0501.2008.01543.x. Epub 2008 May 19. PMID 18492075
- [Background] Lazzara RJ, Porter SS. Platform switching: a new concept in implant dentistry for controlling postrestorative crestal bone levels. Int J Periodontics Restorative Dent. 2006 Feb;26(1):9-17. PMID 16515092
- [Background] Galindo-Moreno P, Leon-Cano A, Monje A, Ortega-Oller I, O'Valle F, Catena A. Abutment height influences the effect of platform switching on peri-implant marginal bone loss. Clin Oral Implants Res. 2016 Feb;27(2):167-73. doi: 10.1111/clr.12554. Epub 2015 Feb 11. PMID 25678247
- [Background] Souza AB, Alshihri A, Kammerer PW, Araujo MG, Gallucci GO. Histological and micro-CT analysis of peri-implant soft and hard tissue healing on implants with different healing abutments configurations. Clin Oral Implants Res. 2018 Oct;29(10):1007-1015. doi: 10.1111/clr.13367. Epub 2018 Sep 23. PMID 30246409
- [Background] Lambrechts T, Doornewaard R, De Bruyckere T, Matthijs L, Deschepper E, Cosyn J. A multicenter cohort study on the association of the one-abutment one-time concept with marginal bone loss around bone level implants. Clin Oral Implants Res. 2021 Feb;32(2):192-202. doi: 10.1111/clr.13689. Epub 2020 Dec 20. PMID 33226676
- [Background] Hamudi N, Barnea E, Weinberg E, Laviv A, Mijiritsky E, Matalon S, Chaushu L, Kolerman R. The Association of the One-Abutment at One-Time Concept with Marginal Bone Loss around the SLA and Platform Switch and Conical Abutment Implants. J Clin Med. 2021 Dec 24;11(1):74. doi: 10.3390/jcm11010074. PMID 35011814
- [Background] Jiang J, Yang H, Zhu H, Bouhamed IEK, Shen X, Lu H, He F. Clinical efficacy of a two-piece abutment conforming to the concept of one abutment one time in the posterior region: A clinical pilot study. Clin Implant Dent Relat Res. 2024 Aug;26(4):763-776. doi: 10.1111/cid.13349. Epub 2024 Jun 6. PMID 38842070
- [Background] Calatrava J, Sanz-Sanchez I, Molina A, Bollain J, Martin C, Sanz M. Effect of one-time placement of the definitive abutment versus multiple healing abutment disconnections and reconnections during the prosthetic phase on radiographic and clinical outcomes: A 12-month randomized clinical trial. Clin Implant Dent Relat Res. 2024 Oct;26(5):998-1011. doi: 10.1111/cid.13361. Epub 2024 Jul 16. PMID 39011816
- [Background] Praca LFG, Teixeira RC, Rego RO. Influence of abutment disconnection on peri-implant marginal bone loss: A randomized clinical trial. Clin Oral Implants Res. 2020 Apr;31(4):341-351. doi: 10.1111/clr.13572. Epub 2020 Jan 27. PMID 31925984
- [Background] Rios-Santos JV, Tello-Gonzalez G, Lazaro-Calvo P, Gil Mur FJ, Rios-Carrasco B, Fernandez-Palacin A, Herrero-Climent M. One Abutment One Time: A Multicenter, Prospective, Controlled, Randomized Study. Int J Environ Res Public Health. 2020 Dec 17;17(24):9453. doi: 10.3390/ijerph17249453. PMID 33348644
- [Background] Moreira F, Rocha S, Caramelo F, Tondela JP. One-Abutment One-Time Effect on Peri-Implant Marginal Bone: A Prospective, Controlled, Randomized, Double-Blind Study. Materials (Basel). 2021 Jul 27;14(15):4179. doi: 10.3390/ma14154179. PMID 34361372
- [Background] Sanz-Sanchez I, Molina A, Martin C, Bollain J, Calatrava J, Sanz M. The effect of one-time abutment placement on clinical and radiographic outcomes: A 5-year randomized clinical trial. Clin Oral Implants Res. 2024 Jun;35(6):609-620. doi: 10.1111/clr.14256. Epub 2024 Mar 20. PMID 38506392
- [Background] Canullo L, Tallarico M, Gracis S, Vela X, Rodriguez X, Covani U. Clinical Considerations on Strategies That Avoid Multiple Connections and Disconnections of Implant Abutments. Int J Periodontics Restorative Dent. 2020 Jan/Feb;40(1):9-17. doi: 10.11607/prd.3642. PMID 31815968
- [Background] Pommer B, Danzinger M, Leite Aiquel L, Pitta J, Haas R. Long-term outcomes of maxillary single-tooth implants in relation to timing protocols of implant placement and loading: Systematic review and meta-analysis. Clin Oral Implants Res. 2021 Oct;32 Suppl 21:56-66. doi: 10.1111/clr.13838. PMID 34642986
- [Background] Vatenas I, Linkevicius T. One abutment one time vs. repeatable abutment disconnections in implants, restored with cemented / screw retained fixed partial dentures: Marginal bone level changes. A systematic review and meta-analysis. Stomatologija. 2021;23(2):35-40. PMID 34528906
- [Background] Kang Y, Zheng X, Zhang D, Li S, Xu S, Chen L, Zhang Z, Lin X. One-Abutment at One-Time in Posterior Edentulism: A Systematic Review and Meta-Analysis. J Craniofac Surg. 2023 Nov-Dec 01;34(8):e720-e724. doi: 10.1097/SCS.0000000000009428. Epub 2023 May 29. PMID 37253247
- [Background] Koutouzis T, Gholami F, Reynolds J, Lundgren T, Kotsakis GA. Abutment Disconnection/Reconnection Affects Peri-implant Marginal Bone Levels: A Meta-Analysis. Int J Oral Maxillofac Implants. 2017 May/June;32(3):575-581. doi: 10.11607/jomi.5367. Epub 2017 Mar 23. PMID 28334059
- [Background] Tallarico M, Caneva M, Meloni SM, Xhanari E, Covani U, Canullo L. Definitive Abutments Placed at Implant Insertion and Never Removed: Is It an Effective Approach? A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Oral Maxillofac Surg. 2018 Feb;76(2):316-324. doi: 10.1016/j.joms.2017.08.025. Epub 2017 Aug 24. PMID 28923270
- [Background] de Carvalho Barbara JG, Luz D, Vianna K, Porto Barboza E. The influence of abutment disconnections on peri-implant marginal bone: A systematic review. Int J Oral Implantol (Berl). 2019;12(3):283-296. PMID 31535098
- [Background] De Pascalis F. Soft tissue integration with a hybrid abutment using the "one abutment-one time" therapeutic protocol: case series. Quintessence Int. 2022 Jun 20;53(7):590-596. doi: 10.3290/j.qi.b3082565. PMID 35723484
- [Background] Waltenberger L, Wolfart S. SafetyCrown: a patient-centered, fully digital concept for immediate implant restoration following the one-abutment/one-time concept-a pilot case series of a new treatment concept. Int J Implant Dent. 2022 Sep 6;8(1):35. doi: 10.1186/s40729-022-00434-2. PMID 36068381
- [Background] Reis INRD, Todescan FF, Ruiz GM, da Silva EVF, Romito GA, Spin-Neto R, Pannuti CM. Influence of supracrestal tissue height on peri-implant hard and soft tissues of single implants placed in the esthetic area using the one abutment-one time approach: a 1-year prospective interventional study. Quintessence Int. 2023 Jul 17;54(7):536-547. doi: 10.3290/j.qi.b4009377. PMID 37013667
- [Background] Henao PAR, Queija LC, Linder S, Dard M, Gonzalez AL, Carrion JB. Clinical and Radiographic Outcomes of a New Fully Tapered Implant with the One-Abutment One-Time Approach: In-Line Clinical Case Series with a 1-Year Follow-up. Int J Oral Maxillofac Implants. 2023 Oct 17;38(5):943-953. doi: 10.11607/jomi.10276. PMID 37847836
- [Background] Ibrahim AM, Elgamal M, Ragheb NA. One-time definitive attachment connection versus healing abutment placement for an implant-retained mandibular overdenture: Peri-implant metabolic activity. J Prosthet Dent. 2024 Oct;132(4):782.e1-782.e7. doi: 10.1016/j.prosdent.2024.03.008. Epub 2024 Apr 10. PMID 38600003
- [Background] Wang YM, He JC. [Short-term follow up of treatment effect using one-time one-abutment placement in implant restoration in 35 patients with single posterior teeth loss]. Shanghai Kou Qiang Yi Xue. 2024 Apr;33(2):156-159. Chinese. PMID 39005091

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1. Read, sign, and receive a copy of the consent form.
  2. Male or female, at least 18 years old, with good oral and general health.
  3. Healed edentulous site with two or more missing teeth in the posterior maxilla or mandible (excluding third molars).
  4. Adequate bone width and height for a 4.3 mm diameter, 8 mm length implant.
  5. Have at least 8 mm restorative space.
  6. Willing to participate and attend a 1-year follow-up before implant restoration procedures.
Pre-assignment Details: 19 participants were initially enrolled. 2 participants withdrew: one moved away during the COVID-19 pandemic, and another agreed to participate and signed the consent form but later withdrew due to being unable to attend the scheduled surgery.
Units Other Than Participants: Implants
Groups:
- Control Group: Control group: Healing abutments are connected on the implants on the day of surgery, which will be subjected to multiple disconnections and reconnections during 1 year follow-up before implant restoration procedures.
- Test Group: Test group: Definitive abutments connected to the implants on the day of surgery. No disconnection or reconnection during 1 year follow-up before implant restoration procedures.
Period: Overall Study
Arm/Group | Control Group | Test Group
Started | 19; 20 Implants | 19; 20 Implants
Completed | 17; 19 Implants | 17; 19 Implants
Not Completed | 2; 1 Implants | 2; 1 Implants
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Units Other Than Participants: Implants
Groups:
- Split Mouth Subject: Control group: Healing abutments are connected on the implants on the day of surgery, which will be subjected to multiple disconnection and reconnection during the prosthetic phase
  Test group: Definitive abutments connected to the implants on the day of surgery. No disconnection or reconnection during the prosthetic phase
  Definitive abutment: With two height options available, On1 Base are selected depending on the thickness of the soft tissue. It remains in position from implant placement to finalization, which leaves the soft tissue undisturbed for optimized healing, moved the restorative platform of Nobel Biocare conical connection implants from bone level to tissue level, thereby simplifying the restorative procedures
Arm/Group | Split Mouth Subject
Number analyzed (Participants) | 17
Number analyzed (Implants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Changes in Peri-implant Marginal Bone Level Between Baseline (Implant Placement) and 1 Year Follow up
Description: Standardized digital periapical radiographs were taken at baseline (implant placement) and at the 1-year follow-up using the long-cone paralleling technique with a custom jig. Peri-implant marginal bone levels were measured on both the mesial and distal aspects to assess bone loss. Changes in peri-implant marginal bone levels were calculated by comparing the measurements at the 1-year follow-up to the baseline values.
Time Frame: At baseline (implant placement) and 1 year follow up
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Implants
Groups:
- Control Group: Healing abutments are connected on the implants on the day of surgery, which will be subjected to multiple disconnection and reconnection during the prosthetic phase
- Test Group: Definitive abutments connected to the implants on the day of surgery. No disconnection or reconnection during the prosthetic phase
  Definitive abutment: With two height options available, On1 Base are selected depending on the thickness of the soft tissue. It remains in position from implant placement to finalization, which leaves the soft tissue undisturbed for optimized healing, moved the restorative platform of Nobel Biocare conical connection implants from bone level to tissue level, thereby simplifying the restorative procedures
Arm/Group | Control Group | Test Group
Number analyzed (Participants) | 17 | 17
Number analyzed (Implants) | 19 | 19
millimeters | 0.80 (0.92) | 0.32 (0.47)
Statistical Analysis 1: Comparison: Control Group vs Test Group; The null hypothesis was that there would be no significant difference in peri-implant bone levels between implants with definitive abutments delivered at the time of surgery, and those subjected to multiple abutment disconnections and reconnections. Power analysis was performed and showed that a sample size of 38 implants was needed to achieve 80% power to detect a difference between the null proportion of 0.500 at a significance level of 0.05; Test type: Superiority; p = 0.009, Wilcoxon (Mann-Whitney); The Shapiro-Wilk test assessed data normality, and paired t-tests or Wilcoxon tests were applied based on normality results; Mean Difference (Final Values) = 0.48, 95% CI 2-sided [0.10 to 0.85], Standard Error of Mean 0.18

2. Secondary Outcome: Changes in Keratinized Mucosa Width
Description: The width of the keratinized mucosa was measured at the mid-buccal aspect of the abutments using a periodontal probe with 1.0 mm markings. Measurements were repeated at the 1-year follow-up at the same location and compared to the baseline values.
Time Frame: At baseline (implant placement) and 1 year follow up
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Implants
Arm/Group | Control Group | Test Group
Number analyzed (Participants) | 17 | 17
Number analyzed (Implants) | 19 | 19
millimeters | 0.90 (0.77) | 0.42 (0.42)
Statistical Analysis 1: Comparison: Control Group vs Test Group; The null hypothesis was that there would be no significant difference in peri-implant bone levels between implants with definitive abutments delivered at the time of surgery, and those subjected to multiple abutment disconnections and reconnections. Power analysis was performed and showed that a sample size of 38 implants was needed to achieve 80% power to detect a difference between the null proportion of 0.500 at a significance level of 0.05. Type of Statistical Test; Test type: Superiority; p = 0.049, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.75, 95% CI 2-sided [-0.0000168 to 1.25], Standard Error of Mean 0.23

3. Secondary Outcome: Changes in Lingual Mucosa Thickness
Description: The thickness of the lingual mucosa at each implant site was measured at the center of the implant site from the bone crest using a periodontal probe with 1.0 mm markings. Measurements were repeated at the 1-year follow-up at the same location and compared to the baseline values taken on the day of implant surgery.
Time Frame: At baseline (implant placement) and 1 year follow up
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Implants
Arm/Group | Control Group | Test Group
Number analyzed (Participants) | 17 | 17
Number analyzed (Implants) | 19 | 19
millimeters | 0.71 (0.59) | 0.38 (0.26)
Statistical Analysis 1: Comparison: Control Group vs Test Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.053, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.38, 95% CI 2-sided [-0.0000522 to 0.75], Standard Error of Mean 0.15

4. Secondary Outcome: Implant Success Rate According to the 2017 Classification Criteria Set by the American Academy of Periodontology (AAP)
Description: Success was determined by the implant's ability to meet these clinical factors, such as the absence of pain, infection, mobility, and radiographic bone loss beyond the acceptable threshold of the follow-up period, as assessed at 12 months post-surgical implantation.
Time Frame: 12 months after surgical implantation
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | Control Group | Test Group
Number analyzed (Participants) | 17 | 17
Number analyzed (Implants) | 19 | 19
Implants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Control Group | Test Group
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-10): https://cdn.clinicaltrials.gov/large-docs/86/NCT04043286/Prot_SAP_000.pdf